CLINICAL TRIAL: NCT01842204
Title: Evaluation of the Efficacy of Electromagnetic Therapy on Postoperative Surgical Pain After Uni- and Bilateral Inguinal Hernia Repair.
Acronym: ELEFANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: BioElectronics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/234
Record Dates: First submitted 2013-04-24; First posted 2013-04-29 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Inguinal Hernias
Keywords: inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- active kit (Experimental): Patient receives an active kit with pulsed electromagnetic field over wound surface area.
  Interventions: Device: Magnetic field therapy device
- non-active kit (Placebo Comparator): Patient receives a non-active kit.
  Interventions: Device: Non magnetic field therapy device.

INTERVENTIONS:
Device: Magnetic field therapy device — Therapy device for 1 week.
  Other Names: Post-surgical and wound care recovery kit.
  Arms: active kit
Device: Non magnetic field therapy device. — Non-active device for 1 week.
  Other Names: Post-surgical and Wound care recovery kit.
  Arms: non-active kit

SUMMARY:
A monocentric interventional randomized placebo controlled trial evaluating the efficacy of the post surgical and wound care recovery kit.

It's a small device that consists of a thin metal ring that is placed on the skin surface, non-invasively. It's connected with a small battery. When the plastic tag is removed and the button is pushed the device is activated. Within the ring a Pulsed Electromagnetic Field is created. It influences the receptor-ligand binding at the cell surface and might improve wound healing by diminishing wound edema and inflammation. It possibly helps reducing the inflammatory reaction induced by surgery.

Patients will be treated for uni or bilateral inguinal hernias and at the end of surgery, at the time of bandage, a kit will be applied at the level of the incision. One group will at random receive a working device, the other half will have a kit without active electromagnetic field.

Postoperative analgesic consumption will be measured in a diary and pain and quality of life will be measured using Visual Analogue Scale and EuraHS-Quality Of Life questionnaires.

The aim of this study is to evaluate whether the placement of the device reduces the acute postoperative pain and whether it reduces the incidence of chronic groin pain.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient
* Primary, unilateral and bilateral groin hernias

Exclusion Criteria:

* No written informed consent
* Recurrent hernias
* 'Incarcerated' hernias
* pregnant women: reaction of a Pulsed Electromagnetic Field on the foetus is unknown
* Patients with pacemaker or Internal defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesic requirement after 1 week. | 1 week after the surgery.
  Evaluation through Questionnaires, VAS, euraHS QOL, diary.

SECONDARY OUTCOMES:
chronic pain at 3 months post-surgery. | 3 months post surgery.
  Clinical evaluation and VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, PhD, FACS, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be